CLINICAL TRIAL: NCT06381479
Title: Exploring the Effects of Probiotics on Workplace Related Stress Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chi-Chang Huang, Dean of Research and Development Office, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B031
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Stress; Sleep Disorder
Keywords: probiotics
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics (Experimental): Probiotic capsules
  Interventions: Dietary Supplement: probiotics
- placebo (Placebo Comparator): Placebo capsules
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotics — each capsule contains Lactiplantibacillus plantarum and Lacticaseibacillus paracasei, 2 caps daily use
  Arms: probiotics
Dietary Supplement: placebo — The placebo capsule contains microcrystalline cellulose, 2 caps daily use.
  Arms: placebo

SUMMARY:
There is still a lack of research to explore the interaction between high-pressure workers and probiotics to improve the intestinal microbiota, sleep, inflammation and anti-oxidation. A total of 120 subjects are expected to be recruited and divided into two groups of 60 subjects, receiving probiotics or placebo, and completing a 8-week trial period.

DETAILED DESCRIPTION:
This is a double blind, randomized control study, which will be conducted by National Taiwan Sport University. A total of 120 subjects are expected to be recruited and divided into two groups of 60 subjects, receiving probiotics or placebo, and completing a 8-week trial period. Volunteers will be asked to fill in the Perceived Stress Scale questionnaire before recruiting. Subjects who meet the criteria will be asked to fill the different questionnaires to evaluate their stress, emotions, gastrointestinal tract symptoms, sleep status and blood draw is also needed.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 60 years old
* Perceived Stress Scale (PSS) score is greater than or equal to 14 points

Exclusion Criteria:

* Have used antibiotics or probiotic products in powder, capsule or tablet form within one month
* Those who are taking Chinese medicine or Western medicine to treat severe acute diseases
* Patients with uncontrolled high blood pressure or diabetes, a history of cancer, and mental illness
* Pregnant or breastfeeding
* Those who have participated in other interventional clinical studies in the past three months
* Who has conflict of interest with PI or unsuitable to participate in the research such as students directly supervised by the project host and those who are unable to read the consent form

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Cortisol | From Baseline to 8 Weeks Assessed
  Cortisol is a steroid hormone that is produced by the adrenal glands which sit on top of each kidney. When released into the bloodstream, cortisol can act on many different parts of the body and can help: body respond to stress or danger increase body's metabolism of glucose control blood pressure reduce inflammation. Cortisol is also needed for the fight or flight response which is a healthy, natural response to perceived threats. The amount of cortisol produced is highly regulated by body to ensure the balance is correct.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | From Baseline to 8 Weeks Assessed
  The PSS scores is a rating tool used to gauge the course of stree. The minimum total score possible is 0 and the maximum total score possible is 40. Higher values represent a worse outcome.
Job Stress Scale | From Baseline to 8 Weeks Assessed
  The job stress scale from Ministry of Labor is a rating tool used to gauge of stress.
Overwork Survey | From Baseline to 8 Weeks Assessed
  This survey is used as self-evaluation of whether an employee overworks, based on the Overwork Survey by Occupational Safety and Health Administration, Ministry of Labor. The survey includes personal-related overwork and work-related overwork.
Insomnia Severity index (ISI) | From Baseline to 8 Weeks Assessed
  The ISI is a rating tool used to gauge of sleeping. Higher values represent a worse outcome.The minimum total score possible is 0 and the maximum total score possible is 28. Higher values represent a worse outcome.
The State Trait Anxiety Inventory (STAI) | From Baseline to 8 Weeks Assessed
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Depression Anxiety Stress Scales (DASS-42) | From Baseline to 8 Weeks Assessed
  The measure of stress with stress subscale in magnesium and placebo groups will be performed in order to assess the impact of the dietary supplement on this parameter. This subscale consists of 14 questions of self-evaluation, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of stress
The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16, QLESQ-16 | From Baseline to 8 Weeks Assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 (QLESQ-16) is a valid, reliable self-report instrument for assessing quality of life. The minimum total score possible is 14 and the maximum total score possible is 70. The higher score the better satisfaction.
VAS-GI | From Baseline to 8 Weeks Assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking probiotics.
Patient Global Impression scales of Improvement rated by patient, PGI-C | From Baseline to 8 Weeks Assessed
  The PGIC is a single-item questionnaire that asks the patient to assess their TD symptoms at specific visits after initiating therapy. The PGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy.
Serotonin | From Baseline to 8 Weeks Assessed
  Levels of serotonin in serum
GABA | From Baseline to 8 Weeks Assessed
  Levels of GABA in serum
Norepinephrine | From Baseline to 8 Weeks Assessed
  Levels of Norepinephrine in serum
Immunoglobulin A, IgA | From Baseline to 8 Weeks Assessed
  Levels of Immunoglobulin A, IgA in serum
adrenocorticotropic hormone, ACTH | From Baseline to 8 Weeks Assessed
  Levels of adrenocorticotropic hormone, ACTH in serum
Total Antioxidant Capacity , TAC | From Baseline to 8 Weeks Assessed
  Levels of Total Antioxidant Capacity , TAC in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Institute of Sports Science, National Taiwan Sport University, Taoyuan District, Taiwan